CLINICAL TRIAL: NCT04148443
Title: Impact of Preoxygenation Time on End-tidal Oxygen Concentration and on Hypoxic Events Occurring After Intubation in the Intensive Care Unit.
Acronym: IMPROVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No inclusion after the 2 years of approval of the human subject review, even after 2 years of prorogation
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHRO-2019-11
Record Dates: First submitted 2019-09-05; First posted 2019-11-01 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Preoxygenation; Intubation; Intensive Care Unit
Keywords: preoxygenation; intubation; end-tidal of oxygen concentration; intensive care unit; critically ill patients

STUDY DESIGN:
Intervention Model Description: Pilot study Randomized controlled multicenter trial Ratio 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 minutes period of preoxygenation (Experimental): 3 minutes of preoxygenation : participants in this group will receive 3 minutes of preoxygenation before intubation
  Interventions: Other: Preoxygenation
- 5 minutes period of preoxygenation (Experimental): 5 minutes of preoxygenation: participants in this group will receive 5 minutes of preoxygenation before intubation
  Interventions: Other: Preoxygenation (longer)

INTERVENTIONS:
Other: Preoxygenation — participants will receive 3 minutes of preoxygenation before intubation
  Arms: 3 minutes period of preoxygenation
Other: Preoxygenation (longer) — participants will receive 5 minutes of preoxygenation before intubation
  Arms: 5 minutes period of preoxygenation

SUMMARY:
Preoxygenation is recommended before performing tracheal intubation. In intensive care units (ICU) patients, there is no specific recommendation regarding the duration of preoxygenation, which usually is applied for 3 to 5 minutes. Monitoring the effectiveness of preoxygenation with end-tidal oxygen concentration (EtO2) is strongly recommended in the operating room but it is never used in ICUs. The first aim of this pilot study is to assess the effect of the preoxygenation duration on EtO2, and secondarily, as an exploratory objective, to determine whether targeting a given value of EtO2 during preoxygenation might insure a safer intubation than when targeting pulse oximetry (SpO2).

DETAILED DESCRIPTION:
This is a multicenter randomized controlled pilot study. 110 patients who require intubation in the ICU will be randomly assigned, with a 1:1 ratio, to 3 or 5 minutes of preoxygenation duration. EtO2 will be continuously measured but hidden to the clinician. The primary outcome measure will be the obtention of an optimal preoxygenation defined by an EtO2 >90%. Secondary outcomes include the occurrence of hypoxia and complications during the procedure.

A pulse oximetry (SpO2) greater than or equal to 96% (SpO2 ≥ 96%) at the end of preoxygenation will be the target in each group. If at the end of the preoxygenation, SpO2 is still lower than 96%, clinician will be allowed to extend the duration of preoxygenation (up to 5 minutes in the 3 minutes period of preoxygenation group and up to 8 minutes in the 5 minutes period of preoxygenation group).

End-tidal oxygen concentration (EtO2) will be measured during preoxygenation and will be hidden to the clinician in order to not influence the duration of preoxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Requiring intubation in ICU
* Free express oral and informed consent of the patient or a proxy in case of impossibility for the patient to consent; emergency inclusion possible when legal representatives and patient's family are not present

Exclusion Criteria:

* Intubation for cardiac arrest
* End-tidal oxygen concentration monitoring not available
* Preoxygenation with high-flow nasal oxygenation
* Previous participation to the study
* Patient known, at time of inclusion, as being under guardianship, tutorship or curator
* Pregnancy or breastfeeding
* Lack of social security number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who reach an EtO2 of 90% | 3 minutes
  To compare the percentage of patients who reach an EtO2 of 90% or higher (optimal preoxygenation) at the end of the preoxygenation period between patients randomized in the 3-min and those randomized in the 5-min preoxygenation duration group.

SECONDARY OUTCOMES:
Expired oxygen fraction (FeO2) | end of the preoxygenation period
  FeO2 will be recorded at the end of the preoxygenation period
Incidence of hypoxemia | 5 minutes after intubation
  Hypoxemia will be defined by SpO2<90% during the intubation procedure
Incidence of severe hypoxemia | End of preoxygenation
  Severe hypoxemia will be defined by SpO2<80% for more than 5 seconds during the intubation procedure from the end of preoxygenation to 5 minutes after invasive mechanical ventilation
Incidence of severe complications | 30 minutes after intubation
  Severs complications occuring within 30 minutes following the intubation procedure will be evaluate and compare between the two groups
Lowest Pulsed saturation with Oxygen (SpO2) | 30 minutes after the end of preoxygenation
  The lowest SPO2 obtained within 30 minutes after the end of preoxygenation will be compared between the 2 groups
Expired oxygen fraction (FeO2) | Through preoxygenantion, i.e., an average of 4 minutes (a minimum of 3 and a maximum of 8 minutes)
  FeO2 during preoxygenation will be recorded every minutes
Partial Pressure of Oxygen (PaO2) | 0 minute
  Measurement of PaO2
Partial Pressure of Oxygen | at the 4th minute on average (3rd or 5th minute depending on the randomisation group)
  Measurement of PaO2 at the end of the preoxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Mai-ANh NAY, MD, Principal Investigator — CHR Orléans
Locations (3):
- France (3):
  - CH de DAX, Dax
  - CHR d'Orléans, Orléans
  - CHRU de TOURS, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrillo A, Gonzalez-Diaz G, Ferrer M, Martinez-Quintana ME, Lopez-Martinez A, Llamas N, Alcazar M, Torres A. Non-invasive ventilation in community-acquired pneumonia and severe acute respiratory failure. Intensive Care Med. 2012 Mar;38(3):458-66. doi: 10.1007/s00134-012-2475-6. Epub 2012 Feb 9. PMID 22318634
- [Background] Thille AW, Frat JP, Brun-Buisson C. Trends in use and benefits of non-invasive ventilation as first-line therapy in acute respiratory failure. Intensive Care Med. 2014 Aug;40(8):1179-80. doi: 10.1007/s00134-014-3370-0. Epub 2014 Jun 25. No abstract available. PMID 24962719
- [Background] Ozsancak Ugurlu A, Sidhom SS, Khodabandeh A, Ieong M, Mohr C, Lin DY, Buchwald I, Bahhady I, Wengryn J, Maheshwari V, Hill NS. Use and outcomes of noninvasive positive pressure ventilation in acute care hospitals in Massachusetts. Chest. 2014 May;145(5):964-971. doi: 10.1378/chest.13-1707. PMID 24480997